CLINICAL TRIAL: NCT06915181
Title: Clinical Usefulness and Influence on Esophageal Motility of Pyridostigmine for Dysphagia in Systemic Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistically the study had to be stopped.
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PySyS
Record Dates: First submitted 2023-04-18; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Systemic Sclerosis With Dysphagia
MeSH Terms: interventions — Pyridostigmine Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo first-then Pyridostigmine (Placebo Comparator)
  Interventions: Drug: Pyridostigmine
- Pyridostigmine first-then Placebo (Active Comparator)
  Interventions: Drug: Pyridostigmine

INTERVENTIONS:
Drug: Pyridostigmine — Subjects will participate in a double-blind randomized controlled cross-over trial. All patients will receive the study drug and placebo. Subjects and investigators will remain blinded to whether the subject receives active treatment during the first or second treatment period.
  Participation in the study will last 10 weeks, with 4 weeks on active treatment and 4 weeks on placebo, with a 2-week wash-out period in between.

SUMMARY:
Systemic sclerosis is characterized by progressive fibrosis of different organ systems. With a longer duration, the risk of gastrointestinal involvement increases. There is a high prevalence of gastro-esophageal reflux disease (GERD) secondary to a severe insufficiency of the lower esophageal sphincter (LES), resulting in severe reflux esophagitis when left untreated. On the long run, this is associated with an elevated risk of esophageal bleeding, peptic stenosis, Barrett esophagus and associated risk of esophageal cancer. Apart from the insufficiency of the LES, esophageal aperistalsis is frequently observed. This results in prolonged esophageal contact with the refluxate due to insufficient clearance by the absence of adequate peristalsis. As a consequence of impaired peristalsis, patients with esophageal involvement in systemic sclerosis often experience dysphagia for solids, causing weight loss and malnu-trition, and reducing in quality of life.

To control reflux disease, high dose proton pump inhibitor therapy is part of the advocated treatment for esophageal involvement in systemic sclerosis. This therapy is highly effective in reducing acidic reflux, but has no influence on the esophageal motility disorder, leaving the dysphagia untreated. Because of the lack of a specific treatment targeting dysphagia, most patients eventually are advised to take conservative measures such as eating while sitting up straight, chewing well and flushing every food bolus with fluids.

While current treatment targets the acidic reflux, there is no accepted treatment to improve esophageal motility. In the presence of dysphagia patients are advocated to follow conservative measures like sitting upright when eating and drinking water to help passage of the bolus.

A cholinesterase inhibitor, pyridostigmine prevents the degradation of acetyl choline at the neuromuscular junction, prolonging its excitatory action. A recent uncontrolled study in patients suffering from systemic sclerosis identified a beneficial effect on gastro-intestinal symptoms, especially constipation. In healthy volunteers intake of pyridostigmine enhanced esophageal contractility as revealed by an increased amplitude of distal esophageal con-tractions. Despite this beneficial influence on esophageal motility there are no data on the possible therapeutic effects in patients with systemic sclerosis and esophageal involvement.

This study aims at evaluating the effects of pyridostigmine on symptoms of dysphagia. Additionally improvement of GERD symptoms and quality of life will be recorded. Improvement of parameters of esophageal motility as well as baseline esophageal impedance during esophageal contraction will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older;
* Known systemic sclerosis;
* Dysphagia with BEDQ score of 10 or more despite twice daily high dose PPI (omeprazole 40 mg b.i.d., esomeprazole 20 mg b.i.d., pantoprazole 40 mg b.i.d., lansoprazole 30 mg b.i.d.).

Exclusion Criteria:

* Presence of reflux oesophagitis grade C or more, eosinophilic oesophagitis, oesophageal stenosis (whether peptic or malignant);
* Prior oesophageal surgery, endoscopic resections, Radiofrequency Abla-tion for Barrett's mucosa or POEM;
* Prior gastric surgery;
* Prior diagnosis of major oesophageal motor disorder such as oesophageal spasm, achalasia, EGJ outflow obstruction;

Prevention of major side effects by exclusion of certain patient groups

* Diarrhoea (defined as Bristol Stool Scale > 5) for more than 2 days per week in the past 2 weeks;
* Uncontrolled asthma, exacerbation of COPD in the last 4 weeks;
* Known ischaemic heart condition or myocardial infarction in the last 4 weeks;
* Resting heart rate < 60 bpm;
* AV-block 2 or 3 (except after implantation of a pacemaker), or bradycardia < 60 bpm;
* Systolic blood pressure > 100 mmHg;
* Impaired renal function with glomerular filtration rate < 30 ml/min;
* Prior or current urinary obstruction;
* Previous treatment with pyridostigmine in the past 4 weeks;
* Treatment with anticholinergic agents in the past 4 weeks;
* Treatment with prokinetic agents during the past 4 weeks
* Pregnancy. Women of childbearing age will undergo a pregnancy test be-fore starting treatment and will be required to use at least 2 highly effective anticonception methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
difference in FSSG score | from baseline till visit 4 (week 10)
  decrease in FSSG score between treatment arms

SECONDARY OUTCOMES:
difference in BEDQ score | from baseline till visit 4 (week 10)
  decrease in BEDQ score between treatment arms
change in quality of life between treatment arms | from baseline till visit 4 (week 10)
  change in quality of life assessed by SF-36 between treatment arms
changes in high resolution manometry between treatment arms | from baseline till visit 4 (week 10)
  differences between mean distal contractility integral
changes in high resolution manometry between treatment arms | from baseline till visit 4 (week 10)
  differences between mean distal latency
changes in high resolution manometry between treatment arms | from baseline till visit 4 (week 10)
  differences between resting pressure of the lower oesophageal sphincter
changes in high resolution manometry between treatment arms | from baseline till visit 4 (week 10)
  differences between percentage of succesful bolus clearance
changes in high resolution manometry between treatment arms | from baseline till visit 4 (week 10)
  differences between percentage of normal peristalsis
changes in oesophageal baseline impedance between treatment arms | from baseline till visit 4 (week 10)
  differences between oesophageal contraction